CLINICAL TRIAL: NCT03887429
Title: An Exploratory, Placebo-Controlled, Crossover Study to Examine the Safety and Activity of SXC-2023 to Improve Behavioral Dynamics in Non-Treatment Seeking Adults Undergoing Acute Nicotine Withdrawal
Brief Title: Restoring Cognitive Control (ReCon) in Acute Nicotine Withdrawal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Promentis Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-202
Record Dates: First submitted 2019-03-14; First posted 2019-03-25 (Actual); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Impulse Control Disorders
Keywords: SXC-2023; Cognitive Control; Impulsivity; Delay Aversion; Top Down Processing; Behavioral Addiction
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SXC-2023 200 mg followed by placebo (Experimental): SXC-2023 200mg dosed once daily for 5 days, followed by 9 day washout, then Placebo dosed once daily for 5 days.
  Interventions: Drug: SXC-2023; Drug: Placebos
- Placebo followed by SXC-2023 200 mg (Experimental): Placebo dosed once daily for 5 days, followed by 9 day washout, then SXC-2023 200mg dosed once daily for 5 days.
  Interventions: Drug: SXC-2023; Drug: Placebos
- SXC-2023 800 mg followed by placebo (Experimental): SXC-2023 800mg dosed once daily for 5 days, followed by 9 day washout, then Placebo dosed once daily for 5 days.
  Interventions: Drug: SXC-2023; Drug: Placebos
- Placebo followed by SXC-2023 800 mg (Experimental): Placebo dosed once daily for 5 days, followed by 9 day washout, then SXC-2023 800mg dosed once daily for 5 days.
  Interventions: Drug: SXC-2023; Drug: Placebos

INTERVENTIONS:
Drug: SXC-2023 — SXC-2023 oral capsules
Drug: Placebos — Matching Placebo oral capsules

SUMMARY:
The purpose of this study is to explore the safety, tolerability and activity of SXC-2023 or placebo when dosed for 5 days in adults with tobacco use disorder who voluntarily abstain from the use of cigarettes.

DETAILED DESCRIPTION:
This study is a Phase 2A, randomized, double-blinded, placebo-controlled, two-period crossover study to evaluate the effect of two doses of SXC-2023 on measures of impulsivity and inhibitory control, urge for cigarettes, and mood in non-treatment seeking smokers who are abstaining from smoking. The study consists of a screening period of up to 30 days, a 5 day randomized double-blind treatment period, a 9 day washout period, followed by a second 5 day randomized double-blind treatment period, with a safety follow-up period 7 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, female or male, 28-55 years of age, inclusive at screening.
2. BMI ≥ 16.0 and ≤ 35.0 kg/m2 at screening.
3. Has provided signed written informed consent and has willingness and ability to comply with all aspects of the protocol, including abstaining from the use of tobacco/nicotine products for two 5-day periods.
4. Non-treatment seeking smokers regularly using tobacco with a FTND score ≥4 at screening and self-reported use of ≥10 cigarettes/day at screening.
5. Has smoked for >5 years at screening.
6. Meets Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria for tobacco use disorder.
7. Must have a score ≥ 4 on the FTND and an expired-air CO level ≥10 ppm during initial screening and prior to first dose.
8. For a female of childbearing potential: either be sexually inactive (abstinent as a life style) for 28 days prior to the first dosing and throughout the study or be using one of the following acceptable birth control methods:

   * Oral contraceptives used for at least 3 months prior to the first dose.
   * Non-hormone releasing intrauterine device for at least 3 months prior to the first dose and with either a physical (e.g., condom, diaphragm, or other) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study.
   * Double physical barrier method (e.g., condom and diaphragm) from 14 days prior to the first dose and throughout the study.
9. Female of non-childbearing potential: must have undergone one of the following sterilization procedures, at least 6 months prior to the first dose:

   1. hysteroscopic sterilization;
   2. bilateral tubal ligation or bilateral salpingectomy;
   3. hysterectomy;
   4. bilateral oophorectomy; Or be postmenopausal with amenorrhea for at least 1 year prior to the first dose with serum follicle stimulating hormone levels consistent with postmenopausal status or have medically documented history of biological or congenital sterility.
10. Has not used Aricept 30 days prior to screening.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems or clinically significant abnormality at the time of the screening visit or expected during the conduct of the study.
2. Subject suffered a concussion 6 months or less prior to screening.
3. Females who are pregnant or breastfeeding.
4. Positive for active hepatitis, human immunodeficiency virus (HIV), coagulopathy, or hepatic illness.
5. Use of Selective Serotonin or Norepinephrine Reuptake Inhibitors for psychiatric illness (e.g. depression, anxiety, etc.), unless subject has been on a stable dose for at least 30 days prior to screening.
6. Use of antipsychotics or use of antiepileptics within 30 days prior to screening.
7. Use of NAC within 30 days prior to screening.
8. Use of Chantix or related smoking cessation medications (e.g., NicoDerm patch, Nicorette gum, etc) within 30 days prior to the first dose.
9. Use of sulfasalazine (Azulfidine®) within 30 days prior to the first dose.
10. DSM-5 criteria for alcohol/substance use disorder (except for tobacco use disorder).
11. History or presence of clinically significant psychiatric condition (except for tobacco use disorder) or disease in the opinion of the PI or designee.
12. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
13. History of seizures.
14. Any history of psychiatric hospitalization in the past year.
15. Currently participating in a clinical study.
16. Previously participated in any Phase 1 Promentis studies or dosed in this Phase 2A study.
17. FTND score <4 and expelled CO levels <10 ppm at screening and prior to first dose.
18. Any clinically significant laboratory, ECG and/or vital sign abnormalities at screening.
19. Unable to read/understand/speak English.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Celerion Inc., Lincoln, Nebraska
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SXC-2023 200 mg Followed by Placebo | Placebo Followed by SXC-2023 200 mg | SXC-2023 800 mg Followed by Placebo | Placebo Followed by SXC-2023 800 mg
Started | 8 | 9 | 9 | 8
Completed First Intervention (5 Days) | 7 | 8 | 7 | 7
Completed Washout (9 Days) | 7 | 8 | 7 | 7
Completed Second Intervention (5 Days) | 7 | 8 | 7 | 7
Completed | 7 | 8 | 7 | 7
Not Completed | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SXC-2023 200 mg Followed by Placebo | Placebo Followed by SXC-2023 200 mg | SXC-2023 800 mg Followed by Placebo | Placebo Followed by SXC-2023 800 mg | Total
Number analyzed (Participants) | 8 | 9 | 9 | 8 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 9 | 8 | 34
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (7.1) | 44 (8.5) | 39 (7.7) | 41 (9.5) | 42 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 4 | 18
  Male | 4 | 4 | 4 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 9 | 8 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 3 | 1 | 3 | 9
  White | 6 | 6 | 6 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 9 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of SXC-2023.
Description: Endpoint assessed using the frequency of serious adverse events, adverse events leading to discontinuation, and adverse events judged to be related to study medication.
Time Frame: Up to 5 days
Measure: Number; unit: Events
Groups:
- During 200 mg SXC-2023 Treatment: AEs observed during treatment with SXC-2023 200 mg.
- During 800 mg SXC-2023 Treatment: AEs observed during treatment with SXC-2023 800 mg.
- During Placebo Treatment: AEs observed during treatment with Placebo.
Arm/Group | During 200 mg SXC-2023 Treatment | During 800 mg SXC-2023 Treatment | During Placebo Treatment
Number analyzed (Participants) | 16 | 16 | 31
Events
  SAEs | 0 | 0 | 0
  AEs leading to study discontinuation | 0 | 0 | 0
  AEs judged to be related to study drug. | 3 | 1 | 12

2. Primary Outcome: Activity of SXC-2023 on Impulsivity, Measured Using Stop Signal Task.
Description: Stop Signal Reaction Time (SSRT) assesses the length of reaction time between a 'go' stimulus and a 'stop' stimulus at which the subject is able to inhibit their motor response 50% of the time. The scale is from 0-1500 milliseconds with a lower value showing reduced motor impulsivity. Subject scores were collected pre-dose on day 1 of treatment and post-dose on day 5 of treatment, and the change in subject scores was assessed.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- SXC-2023 200mg: Change in subjects treated with 200 mg SXC-2023 for 5 days.
- SXC-2023 800mg: Change in subjects treated with 800 mg SXC-2023 for 5 days.
- Placebo: Change in subjects treated with Placebo for 5 days.
Arm/Group | SXC-2023 200mg | SXC-2023 800mg | Placebo
Number analyzed (Participants) | 9 | 8 | 17
milliseconds | 4.6901 (6.7368) | -1.757 (6.8491) | 3.956 (3.9661)
Statistical Analysis 1: Comparison: SXC-2023 800mg vs Placebo; It was hypothesized that treatment with SXC-2023 would reduce impulsivity as measured by SSRT in chronic cigarette smokers abstaining from nicotine for 5 days; Test type: Superiority; p = .009, t-test, 1 sided

3. Primary Outcome: Activity of SXC-2023 on Risk Taking Behavior, as Measured Using Cambridge Gamblers Task - Delay Aversion Total.
Description: Cambridge Gamblers Task measures risk taking behavior using a score from -1 to 1, with a higher value showing increased impulsivity. Subject scores were collected pre-dose on day 1 of treatment and post-dose on day 5 of treatment and change in score assessed.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SXC-2023 200mg | SXC-2023 800mg | Placebo
Number analyzed (Participants) | 9 | 8 | 17
units on a scale | .03236 (.02652) | .01358 (.02655) | .03931 (.01569)
Statistical Analysis 1: Comparison: Placebo; It was hypothesized that 5 days of nicotine abstinence in chronic cigarette smokers would result in increased risk taking behavior as measured using DAVT in subjects receiving placebo as treatment; Test type: Superiority; p = .015, t-test, 1 sided
Statistical Analysis 2: Comparison: SXC-2023 800mg; It was hypothesized that 5 days of nicotine abstinence in chronic cigarette smokers would not result in increased risk taking behavior as measured using DAVT in subjects treated with SXC-2023; Test type: Superiority; p > .1, t-test, 1 sided

4. Primary Outcome: Activity of SXC-2023 on Abstinence Induced Mood, Assessed by Positive and Negative Affect Schedule.
Description: Outcome to be measured using two scores ranging from 10-50, with a higher score indicating a more positive affect, and a lower score indicating a more negative affect. Subject scores were collected pre-dose on day 1 of treatment and post-dose on day 5 of treatment.
Time Frame: Up to 5 days.
Population: Subjects who did not complete treatment with both placebo and SXC-2023 were excluded from analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 200 mg SXC-2023 or Placebo QD: Change in Positive and Negative affect in subjects treated with 200 mg SXC-2023 or placebo for 5 days.
- 800 mg SXC-2023 or Placebo QD: Change in Positive and Negative affect in subjects treated with 800 mg SXC-2023 or placebo for 5 days.
Arm/Group | 200 mg SXC-2023 or Placebo QD | 800 mg SXC-2023 or Placebo QD
Number analyzed (Participants) | 14 | 14
score on a scale
  SXC-2023 Change in Positive Aspect | 3.5 (8.2) | 2.1 (7.0)
  Placebo Change in Positive Aspect | 2.0 (7.43) | 3.3 (6.5)
  SXC-2023 Change in Negative Aspect | -.9 (5.01) | -1.2 (2.61)
  Placebo Change in Negative Aspect | -.7 (3.93) | .1 (5.02)

5. Primary Outcome: Activity of SXC-2023 on Measures of Abstinence Induced Urge for Cigarettes, Assessed by Questionnaire on Smoking Urges.
Description: Outcome to be measured using a score ranging from 10-70, with a higher score indicating a higher urge for a cigarette. Subject scores were collected pre-dose on day 1 of treatment and post-dose on day 5 of treatment.
Time Frame: Up to 5 days.
Population: Subjects who did not complete treatment with both placebo and SXC-2023 were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 200 mg SXC-2023 or Placebo QD: Change in subjects treated with 200 mg SXC-2023 or placebo for 5 days.
- 800 mg SXC-2023 or Placebo QD: Change in subjects treated with 800 mg SXC-2023 or placebo for 5 days.
Arm/Group | 200 mg SXC-2023 or Placebo QD | 800 mg SXC-2023 or Placebo QD
Number analyzed (Participants) | 14 | 14
units on a scale
  SXC-2023 Change in Anticipation of Pleasure | -.3 (1.155) | .64 (1.332)
  Placebo change in Anticipation of Pleasure | -.04 (1.1236) | .17 (.848)
  SXC-2023 change in Anticipation of Relief | .14 (1.201) | .21 (1.214)
  Placebo change in Anticipation of Relief | -.06 (.946) | .46 (.794)

6. Primary Outcome: Activity of SXC-2023 on Measures of Abstinence Induced Urge for Cigarettes, Assessed by Cigarette Evaluation Questionnaire.
Description: Outcome to be measured using five scores ranging from 1-7 and corresponding to "Smoking Satisfaction," "Psychological Reward," "Aversion," "Enjoyment of Respiratory Tract Sensations" and "Craving Reduction." A higher score indicates a greater intensity of the associated sensation. Subject scores were collected pre-dose on day 1 of treatment and post-dose on day 5 of treatment.
Time Frame: Up to 5 days.
Population: Complications with application of scales prevented collection of data from the majority of subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 200 mg SXC-2023 or Placebo QD | 800 mg SXC-2023 or Placebo QD
Number analyzed (Participants) | 5 | 4
units on a scale
  SXC-2023 change in Satisfaction: number analyzed (Participants) | 5 | 3
  SXC-2023 change in Satisfaction | .1 (1.28) | .4 (.51)
  Placebo change in Satisfaction: number analyzed (Participants) | 3 | 4
  Placebo change in Satisfaction | .3 (.33) | -.2 (.69)
  SXC-2023 change in Psychological reward: number analyzed (Participants) | 5 | 3
  SXC-2023 change in Psychological reward | .16 (1.315) | .33 (.808)
  Placebo change in Psychological reward: number analyzed (Participants) | 3 | 4
  Placebo change in Psychological reward | .8 (.693) | -.2 (1.071)
  SXC-2023 change in Aversion: number analyzed (Participants) | 5 | 3
  SXC-2023 change in Aversion | .7 (1.396) | 0 (0)
  Placebo change in Aversion: number analyzed (Participants) | 3 | 4
  Placebo change in Aversion | 0 (0) | .63 (.946)
  SXC-2023 change in Enjoyment of Sensation: number analyzed (Participants) | 5 | 3
  SXC-2023 change in Enjoyment of Sensation | 0 (1.58) | 1.3 (1.53)
  Placebo change in Enjoyment of Sensation: number analyzed (Participants) | 3 | 4
  Placebo change in Enjoyment of Sensation | 0 (2) | .8 (.96)
  SXC-2023 change in Craving Reduction: number analyzed (Participants) | 5 | 3
  SXC-2023 change in Craving Reduction | -.4 (1.14) | .3 (.58)
  Placebo change in Craving Reduction: number analyzed (Participants) | 3 | 4
  Placebo change in Craving Reduction | -.7 (2.08) | 0 (1.41)

7. Primary Outcome: Activity of SXC-2023 on Measures of Abstinence Induced Urge for Cigarettes and Mood, Assessed by Cue Reactivity and Likert Assessment.
Description: Outcome to be measured using two scores, the first ranging from 10-70, with a higher score indicating a stronger urge to smoke, and the second score ranging from 10-80, with a higher score indicating a more positive mood. Subject scores were collected pre-dose on day 1 of treatment and post-dose on day 5 of treatment.
Time Frame: Up to 5 days.
Population: Subjects who did not complete treatment with both placebo and SXC-2023 were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 200 mg SXC-2023 or Placebo QD | 800 mg SXC-2023 or Placebo QD
Number analyzed (Participants) | 14 | 13
units on a scale
  SXC-2023 change in Neutral Urge: number analyzed (Participants) | 13 | 13
  SXC-2023 change in Neutral Urge | .353 (1.7932) | -.052 (1.8934)
  Placebo change in Neutral Urge: number analyzed (Participants) | 13 | 13
  Placebo change in Neutral Urge | -.142 (1.5071) | -.173 (1.5458)
  SXC-2023 change in Neutral Mood: number analyzed (Participants) | 13 | 13
  SXC-2023 change in Neutral Mood | 1.058 (1.3775) | 1.667 (1.6004)
  Placebo change in Neutral Mood: number analyzed (Participants) | 13 | 13
  Placebo change in Neutral Mood | .602 (1.7237) | 1.192 (1.476)
  SXC-2023 change in Positive Urge | .5 (1.922) | .12 (1.793)
  Placebo change in Positive Urge | -.12 (1.543) | -.04 (1.547)
  SXC-2023 change in Positive Mood: number analyzed (Participants) | 13 | 13
  SXC-2023 change in Positive Mood | 1.23 (1.509) | 1.35 (2.065)
  Placebo change in Positive Mood: number analyzed (Participants) | 13 | 13
  Placebo change in Positive Mood | .73 (1.666) | 1.38 (1.557)
  SXC-2023 change in Smoking Urge | .39 (2.105) | -.23 (1.549)
  Placebo change in Smoking Urge: number analyzed (Participants) | 13 | 13
  Placebo change in Smoking Urge | -.65 (1.864) | -.27 (1.653)
  SXC-2023 change in Smoking Mood: number analyzed (Participants) | 13 | 13
  SXC-2023 change in Smoking Mood | .42 (1.352) | 1.65 (1.796)
  Placebo change in Smoking Mood: number analyzed (Participants) | 13 | 13
  Placebo change in Smoking Mood | .88 (1.431) | 1 (1.339)

8. Other Pre Specified Outcome: Levels of Glutathione (GSH) in Whole Blood Following 5 Days of Tobacco Abstinence.
Description: Levels total and/or reduced of GSH in whole blood will be collected at baseline (prior to dosing on Day 1) and after 5 days of tobacco abstinence (after dosing on Day 5). Subject scores were collected pre-dose on day 1 of treatment and post-dose on day 5 of treatment.
Time Frame: Up to 5 days.
Population: Subjects who did not complete treatment with both placebo and SXC-2023 were excluded from analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 200 mg SXC-2023 or Placebo QD | 800 mg SXC-2023 or Placebo QD
Number analyzed (Participants) | 14 | 14
μg/mL
  SXC-2023 change in GSH concentration | -3.45 (23.318) | -20.6 (73.23)
  Placebo change in GSH concentration | -5.13 (21.826) | -5.12 (23.587)

ADVERSE EVENTS:
Time Frame: 5 day treatment period, and following 9 days.
Arm/Group | During 200 mg SXC-2023 Treatment | During 800 mg SXC-2023 Treatment | During Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/31
Other Adverse Events (participants affected / at risk) | 5/16 | 3/16 | 13/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | During 200 mg SXC-2023 Treatment (N=16) | During 800 mg SXC-2023 Treatment (N=16) | During Placebo Treatment (N=31)
Headache (Nervous system disorders) | 2 | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Defecation Urgency (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Thirst (General disorders) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1
Anger (Psychiatric disorders) | 0 | 1 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lacrimation increase (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03887429/Prot_SAP_001.pdf